CLINICAL TRIAL: NCT04852172
Title: A Phase I/IIA Open-label Dose-Finding Study with Subsequent Double-blind, Placebo-controlled, Randomized Study of L-citrulline in Sickle Cell Disease Presenting to Emergency Department (ED) in Vaso Occlusive Crisis (VOC) in Children, Adolescents and Young Adults (6 to 21 Years)
Brief Title: L-citrulline Injection in Patients Aged 6-21 Years Old with Sickle Cell Disease Presenting with Vaso-Occlusive Crisis (VOC)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Impacted by viraemia resulting in higher than expected admissions
Sponsor: Asklepion Pharmaceuticals, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CIT-SCD-001-01
Record Dates: First submitted 2021-03-18; First posted 2021-04-21 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2023-08

CONDITIONS: Acute Vaso Occlusive Crisis (VOC)
MeSH Terms: interventions — Citrulline; serum P-component; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Open-label Dose-Finding Study with Subsequent Double-blind, Placebo-controlled, Randomized Study of L-citrulline in Sickle Cell Disease Presenting to Emergency Department (ED) in Vaso Occlusive Crisis (VOC) in Children, Adolescents and Young Adults (6 to 21 years).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind placebo controlled (Part 2)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- Arm 1 (L-citrulline) (Active Comparator): 25 mg/kg bolus + 9 mg/kg/hr continuous infusion of L-citrulline for up to 7 hours
  Interventions: Drug: L-citrulline
- Arm 2 (L-citrulline) (Active Comparator): 50 mg/kg bolus + 9 mg/kg/hr continuous infusion of L-citrulline for up to 7 hours
  Interventions: Drug: L-citrulline
- Arm 3 (L-citrulline) (Active Comparator): 100 mg/kg bolus + 9 mg/kg/hr continuous infusion of L-citrulline for up to 7 hours
  Interventions: Drug: L-citrulline
- Arm 4 (L-citrulline) (Active Comparator): 100 mg/kg bolus + 11 mg/kg/hr continuous infusion of L-citrulline for up to 7 hours
  Interventions: Drug: L-citrulline
- Part 2 Arm 1 (L-citrulline) (Active Comparator): Subjects will be randomized to 2 of the doses selected from Part 1 and placebo in a 1:1:1 ratio. L-citrulline will be administered to the active arm.
  Interventions: Drug: L-citrulline
- Part 2 Arm 2 D5 1/2NS (Placebo Comparator): Subjects will be randomized to 2 of the doses selected from Part 1 and placebo in a 1:1:1 ratio.
  Interventions: Other: D5 1/2NS

INTERVENTIONS:
Drug: L-citrulline — L-citrulline is a naturally occurring amino acid. It is produced by, and normally present in, the human body.
  Other Names: L-CIT, CIT
  Arms: Arm 1 (L-citrulline); Arm 2 (L-citrulline); Arm 3 (L-citrulline); Arm 4 (L-citrulline); Part 2 Arm 1 (L-citrulline)
Other: D5 1/2NS — Saline
  Other Names: Saline
  Arms: Part 2 Arm 2 D5 1/2NS

SUMMARY:
The purpose of this study is to determine if intravenous L-citrulline can abrogate an active vaso-occlusive crisis in sickle cell disease, resulting in decreased pain, reduction or elimination of opiate usage, and reduction or elimination of hospital admission. The applicant is developing intravenous L-citrulline (Turnobi™) for treatment of sickle cell disease (SCD). The current development program targets treatment of sickle cell-associated vaso-occlusive crisis (VOC) specifically. The aim of Part 1 is to identify the optimum dose regimens for the Part 2 of the trial which is a double-blind, placebo controlled adaptive 'pick-the-winner' design. This study will allow assignment of more subjects to the better treatment arm/s based on emerging data. The study, initially, will evaluate efficacy and tolerability of incremental doses of intravenous (IV) L-citrulline (Turnobi™) in patients with SCD while receiving standard of care therapy for VOC.

DETAILED DESCRIPTION:
Overall Design:

This is a study in children, adolescents, and young adults (6 to 21 years) with SCD presenting to an emergency department (ED) with VOC. Children below age 6 are likely to be recruited in a subsequent phase, once proof of concept is established on optimized dose regimen. Eligible subjects will have documented SCD. Intravenous L citrulline (Turnobi™) or placebo will be administered in addition to standard of care VOC therapy to children, adolescents, and young adults presenting with SCD VOC - defined as painful episode without other apparent causes of pain and without significant organ dysfunction or signs of systemic infection.

This is a single center study, conducted in 2 parts:

Part 1: This is an open-label, ascending dose part of the study. After obtaining the informed consent/assent, the enrolled subjects will be in the ED for up to 7 hours where L-citrulline will be administered as depicted in the dosing panel below. Each dose will be administered sequentially until 5 subjects per dose cohort are accrued.

Dosing panels in Part 1:

25 mg/kg bolus + 9 mg/kg/hr infusion; 50 mg/kg bolus + 9 mg/kg/hr infusion; 100 mg/kg bolus + 9 mg/kg/hr infusion; 100 mg/kg bolus + 11 mg/kg/hr infusion;

After each panel of 5 have been dosed, response to a dose is determined by the Principal Investigator (PI) with the internal review committee based primarily on analgesic effects assessed by review of Visual Analogue Scale (VAS) score, opioid dosing, and tolerability.

If the dose panel is assessed safe and 3 of 5 subjects in a cohort respond to the treatment, the current dose arm will continue to accrue a total of 10 subjects. If the dose panel is assessed as safe; however, fewer than 3 of the 5 subjects respond, the current dose arm will be stopped, and the subjects will be recruited to the next dosing panel.

Two additional panels of 5 to 10 subjects receiving doses outside these ranges may be accrued at the request of the internal review committee if determined necessary to achieve the study's objectives. As long as supported by emerging data, the subjects in these additional panels may receive a lower or higher bolus injection but no greater than 150 mg/kg bolus and/or a lower or higher infusion dose but no greater than 15 mg/kg/hour. Up to 60 subjects may be enrolled in Part 1 of the study with a likely sample size of approximately 40 subjects.

Part 1 of the study is intended to select up to 2 effective and tolerated dose regimens for Part 2 of the study.

Part 2: The optimal dose regimens (at least1 but probably 2) selected from Part 1 will be analyzed in a randomized, double-blind, placebo-controlled adaptive pick-the-winner design. This will allow assignment of more subjects to the better treatment arm/s based on emerging data. Efficacy will be based primarily on analgesic effect assessed by VAS/opioid dose composite, admission or not, and tolerability based on adverse drug reactions by the internal review committee.

A total of 60 subjects will take part in Part 2. Subjects will be randomized to 2 of the doses selected from Part 1 and placebo in a 1:1:1 ratio. After 30 subjects (10 per treatment arm) have been randomized, an interim analysis will be performed. If the higher dose is providing markedly more pain relief than the lower dose - with no safety issues - then the lower dose will be dropped. Otherwise, if efficacy and safety look similar, the lower dose will be retained, and the higher dose will be dropped. In other words, the most successful active treatment arm will be chosen for further study versus placebo. The internal review committee will be responsible for making this decision. Subsequently, 30 more patients will be randomized in a 1:1 fashion in the remaining 2 study arms (15 patients each). In the unlikely case that the placebo arm demonstrates superior response to both active treatment arms, the interval review committee will recommend discontinuing the study.

If after 30 subjects, it is determined by the internal review committee that 1 of the 2 doses is significantly more effective in subjects with particular characteristics, the less effective L-citrulline dose regimen can be dropped for those subjects, eg, if those with more severe VOC only respond to the higher dose but those with less severe VOC respond equally well to either dose, subjects with severe VOC will be adaptively allocated into a separate stratum and randomized only to the higher dose or placebo.

All subjects in both Part 1 and Part 2 will receive standard of care for analgesia per SCD pain management protocol consistent with the Children's national ED guidance guided individualized care plan irrespective of treatment with study treatment or placebo. The end of the study is defined as the date of the last visit of the last subject in the study or last scheduled procedure the last subject in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Sickle cell disease (all genotypes)
2. Children, adolescents and young adults between ages 6 to 21 years
3. In a steady disease state and not in the midst of any acute complication other than VOC due to sickle cell disease at study entry
4. For female of childbearing potential, a negative urine pregnancy test and using an adequate method of contraception, or denies sexual activity
5. Subjects or parents or legal guardian of the subject who are willing and able to sign and provide consent and assent (where appropriate for the age of the child).

Exclusion Criteria:

1. Current pain lasting >3 days
2. >6 hospital admissions in the prior year
3. History of opioid dependence/substance abuse
4. Has been on a clinical trial of a new therapy for sickle cell disease within the last 3 months
5. Presence of any other complication related to sickle cell disease such as splenic sequestration, hepatic sequestration, stroke, avascular necrosis of the hip/shoulder, acute priapism, renal dysfunction, dactylitis, acute chest syndrome and other major medical conditions or organ dysfunction
6. Severe anemia (hemoglobin <6 g/dL)
7. History of red blood cell transfusion within the last 30 days
8. Systemic steroid therapy within the last 48 hours
9. Pregnancy or lactation (subjects must have a negative urine pregnancy test)
10. Serum creatinine levels:

    1. Age 6 to 13 years >0.9 mg/dL
    2. Age 14 to 17 years >1.0 mg/dL
    3. Age >18 years >1.5 mg/dL
11. Report of fever (>38°C) within last 48 hours
12. Presence of acute chest syndrome, sepsis, bacterial infection, hemodynamic instability
13. Subjects with inability to have parental assent given (ages 6 to 17 years) or consent (ages 18 through 21 years).

    Note: Parents or legal guardians can provide consent for subjects who are unable to provide assent (eg, sleepy or preoccupied by their pain).
14. History of allergic reaction to L-citrulline product
15. Medications that are known to be contra-indicated with use of L-citrulline
16. History of diabetes.
17. Subjects with a baseline prothrombin time International Normalized ratio (INR) >2.0.
18. Received any blood products within 3 weeks of the screening visit.
19. Unreliable venous access
20. The PI considers that the subject will be unable to comply with the study requirements.

Ages: 6 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2021-04-29 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Dose Optimization (Part 1) | Collected from enrollment to end of study over 18 months
  During Part 1 of the study four cohorts will be enrolled. Cohorts will be squentially completed. Each cohort has a different dosing schema.
To determine the how the study medication is processed by the body. | Collected from enrollment to Emergency room Discharge, Approximability 7 Hours
  About 5 milliliters of blood will be collected before study medication is administered and then every 15 minutes to measure how much study drug is in your blood stream. The blood sample collected will be analyzed for Pharmacokinetic parameters Peak of drug in the blood will be measured
To determine the how the study medication is processed by the body. | Collected from enrollment to Emergency room Discharge, Approximability 7 Hours
  About 5 milliliters of blood will be collected before study medication is administered and then every 15 minutes to measure how much study drug is in your blood stream. The blood sample collected will be analyzed for Pharmacokinetic parameters Trough of drug in the blood will be measured
To determine the how the study medication is processed by the body. | Collected from enrollment to Emergency room Discharge, Approximability 7 Hours
  About 5 milliliters of blood will be collected before study medication is administered and then every 15 minutes to measure how much study drug is in your blood stream. The blood sample collected will be analyzed for Pharmacokinetic parameters of steady state concentration (Cmax) of drug in the blood will be measured
To determine the how the study medication is processed by the body. | Collected from enrollment to Emergency room Discharge, Approximability 7 Hours
  About 5 milliliters of blood will be collected before study medication is administered and then every 15 minutes to measure how much study drug is in your blood stream. The blood sample collected will be analyzed for Pharmacokinetic parameters of AUC of drug in the blood will be measured
Change in Visual Analogue Scale (VAS) pain score | Collected from enrollment to end of study over 18 months
  Please note that scale info should be entered in the outcome measure description field: at least 2-point decrease or 30% change in pain intensity VAS or Faces Pain Scale score RANGE from 0 (No pain) to 100 (Maximum Pain) (for subjects 6 to 7 years old) when compared with baseline value; assessed every 15 minutes
Change from baseline in amount of overall opioid use | Collected from enrollment to end of study over 18 months
  Opioid consumption will be recorded from baseline to end of study.
Discharge from ED/hospital within 7 hours | Collected from enrollment to end of study over 18 months
  Time spent in the ED/hospital will be collected
Assessment of safety | Collected from enrollment to end of study over 18 months
  The rate of reported AE analysis and Lab abnormalities for each cohort

SECONDARY OUTCOMES:
Preliminary assessment of pain change measured | Collected from enrollment to end of study (2-Days)
  The standard of care Visual Analog Scale (VAS) pain scale will be administered at baseline then every 15 minutes after the start of study
Preliminary assessment of change of opioid use overall | Collected from enrollment to end of study (30 Days)
  The standard of care will be followed for pain management. the amount of opioids consumed will be collected.
Time to clinical resolution of VOC | Collected from enrollment to end of study (30 Days)
  Time to clinical resolution of VOC depicted by sustained VAS score; assessed every 15 minutes
Duration or length of hospital stay | Collected from enrollment to end of study (30-Days)
  Data collected from the ED visit through day 30 follow-up will look at reoccurrence of admission.

CONTACTS AND LOCATIONS:
Overall Officials: Gurdyal Kalsi, MD, MFPM, Study Director — Asklepion Pharmaceuticals, LLC
Locations (2):
- United States (2):
  - Children's National Hospital, Washington D.C., District of Columbia
  - The University of Mississippi Medical Center, Jackson, Mississippi

IPD SHARING:
Plan to Share IPD: No